CLINICAL TRIAL: NCT01843153
Title: Continuous Versus Intermittent Sciatic Block Combined With a Continuous Femoral Block for Patients Undergoing Total Knee Arthroplasty: a Prospective, Randomized Trial.
Brief Title: Continuous Versus Intermittent Sciatic Block for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kreiskrankenhaus Dormagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sciatic block
Record Dates: First submitted 2013-04-25; First posted 2013-04-30 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2013-04

CONDITIONS: Total Knee Arthroplasty; Pain
Keywords: pain score
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intermittent (Other): injection of ropivacaine on demand
  Interventions: Drug: Ropivacaine
- continuous (Other): continuous ropivacaine infusion
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine

SUMMARY:
The role of a sciatic block in addition to a femoral block remains controversial. The study addresses this topic by comparing a continuous block versus an injection on demand.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total knee arthroplasty

Exclusion Criteria:

* failure to establish femoral and sciatic block
* insufficient analgesic effect of the block
* patient declines to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
pain score (VRS) | 4 days

SECONDARY OUTCOMES:
frequency of injections into the sciatic catheter | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- KKH Dormagen, Dormagen, Germany

REFERENCES:
- [Derived] Soltesz S, Meiger D, Milles-Thieme S, Saxler G, Ziegeler S. Intermittent versus continuous sciatic block combined with femoral block for patients undergoing knee arthroplasty. A randomized controlled trial. Int Orthop. 2016 Sep;40(9):1861-7. doi: 10.1007/s00264-016-3117-3. Epub 2016 Jan 25. PMID 26810904